CLINICAL TRIAL: NCT05434585
Title: A Randomized, Double-Blind, and Placebo-Controlled Phase 1 Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Variant mRNA Vaccines (ABO1009-DP and ABO-CoV.617.2) in Indonesian Subjects Aged 18 Years and Older Who Have Not Received SARS-CoV-2 Vaccines
Brief Title: A Study to Evaluate Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Variant (COVID-19) mRNA Vaccines
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABO1009-CoV.617.2-101Indonesia
Record Dates: First submitted 2022-06-20; First posted 2022-06-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: Delta; Omicron; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 60 subjects will be randomized in a 2:2:1 ratio to receive ABO1009-DP, ABO-CoV.617.2, or placebo
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1: ABO1009-DP (Experimental): Intramuscularly injecting 15 μg of ABO1009-DP into lateral deltoid of the upper arm of subjects on D0 and D28, respectively.
  Interventions: Biological: ABO1009-DP
- Test group 2: ABO-CoV.617.2 (Experimental): Intramuscularly injecting 15 μg of ABO-CoV.617.2 into lateral deltoid of the upper arm of subjects on D0 and D28, respectively.
  Interventions: Biological: ABO-CoV.617.2
- Control group: Placebo (Placebo Comparator): Intramuscularly injecting placebo into lateral deltoid of the upper arm of subjects on D0 and D28, respectively
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ABO1009-DP — Vaccine
  Arms: Test group 1: ABO1009-DP
Biological: ABO-CoV.617.2 — Vaccine
  Arms: Test group 2: ABO-CoV.617.2
Other: Placebo — Placebo
  Arms: Control group: Placebo

SUMMARY:
A Phase 1 study to evaluate safety, tolerability, and immunogenicity of SARS-CoV-2 variant mRNA vaccines which are used to prevent COVID-19 caused by SARS-CoV-2 infection. this study is conducted during Indonesian subjects aged 18 years and older who have not received SARS-CoV-2 vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the ICF approved by the Ethics Committee before any study procedure and agree to participate in the study.
2. Healthy male or female able to provide legal identity certificate and aged 18 years and older when signing the ICF.
3. Have not previously received any SARS-CoV-2 vaccine (marketed or investigational) before screening.
4. Be able to communicate well with the investigator, and to understand and comply with the requirements of this clinical trial.
5. Males or females of childbearing potential voluntarily take effective contraceptive methods from signing ICF to 3 months after the last vaccination, including sexual abstinence or effective contraceptive measures (e.g., intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, intrauterine device [IUD], condoms [male], diaphragm, and cervical cap).

Exclusion Criteria:

Exclusion criteria for the first dose

Subjects should not participate in this clinical study if any of the following criteria is met:

1. Subjects who do not meet health standard upon comprehensive physical examination, mainly including:

1. Abnormal vital signs (pulse < 60 bpm or > 100 bpm, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg when keeping awake) with clinical significance.
2. Body mass index (BMI) < 18 kg/m2 or > 30 kg/m2.
3. Abnormal laboratory values and with clinical significance at the investigator's discretion at screening.
4. Subjects who do not remain overall healthy (i.e., is anticipated to have fatal outcome of uncontrolled diseases within 12 months and is not able to provide blood as specified by the trial with anticipated, deleterious medical consequences) in the clinical judgment of the investigator based on medical history and physical examination.

2. SARS-CoV-2 specific antibody positive at screening. 3. Positive SARS-CoV-2 RT-PCR result at screening. 4. Prior medical history of SARS-CoV-2, severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS), or other human coronavirus infections or diseases.

5. Fever (axillary temperature ≥ 37.3℃) on the day of vaccination with this study vaccine or within recent 72 hours.

6. Pregnant or lactating women, or those who plan to donate sperm or egg during the trial.

7. Prior history of allergic reaction or anaphylaxis to any vaccine or its excipients, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc.

8. Prior use of any vaccine within 28 days before using this study vaccine or planning to use any vaccine other than this study vaccine during the study period.

Note: The exception is that licensed influenza vaccines can be received more than 28 days after the second dose of study injection.

9. Participation in the studies of any other interventional device or drug within 30 days before the screening, or current treatment with other investigational drug(s) or within 5 half-lives after taking the last dose of the study drug.

10. Hereditary hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorder), or a history of serious bleeding, or a history of massive bleeding after intramuscular injection or intravenous puncture or ecchymosis.

11. Known medical history or diagnosis confirming that subjects have diseases affecting immune system function, including cancer (except skin basal cell carcinoma), congenital or acquired immunodeficiency (e.g., infection with human immunodeficiency virus [HIV]), uncontrolled autoimmune disease.

12. Serious or uncontrolled respiratory system disorders, cardiovascular disorders, nervous system disorders, blood and lymphatic system disorders, liver and kidney disorders, metabolism and skeletal disorders, etc. influencing study results evaluation at the investigator's discretion.

13. Asplenia or functional asplenia. 14. Long-term use (continuous use ≥ 14 days) of immunosuppressants or other immunomodulators (e.g., glucocorticoids: prednisone or similar drugs) within 6 months prior to administration of this investigational vaccine, except for topical medications (e.g., ointments, eye drops, inhalants or nasal sprays). And the topical medications should not exceed the recommended dose in the labels for use or induce any signs of systemic exposure.

15. Having received immunoglobulins and/or blood products within 3 months prior to administration of this investigational vaccine.

16. Suspected or known alcohol dependency or drug abuse, which may affect safety evaluation or subject's compliance at the investigator's discretion.

17. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits.

18. Receiving antituberculosis treatment. 19. Staff of test site, sponsor and contract research organization (CRO) taking part in the study.

Exclusion Criteria for the second dose

If the subjects have any of the followings prior to the second dose, vaccination will be terminated. However, other study procedures can be continued at the discretion of the investigators:

1. Positive pregnancy test for female subjects of childbearing potential.
2. Positive SARS-CoV-2 RT-PCR result.
3. Serious hypersensitivity or serious adverse event causally related to vaccination has occurred following the first dose.
4. Other circumstances considered by the investigator as inappropriate to receive the second dose of the vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited adverse events (AEs) | 0 to 7 days after each injection
  Solicited adverse events 0 to 7 days after each injection；
Incidence of unsolicited AEs | 0 to 28 days after each injection
  Unsolicited adverse events 0 to 28 days after each injection ； Adverse reactions/events related to blood chemistry, blood routine, blood coagulation function and urinalysis indicators 4 days after each injection
Changes of blood chemistry, blood routine, blood coagulation function and urinalysis indicators 4 days after each injection in comparison to pre-injection | 4 days after each injection in comparison to pre-injection
  Adverse reactions/events related to blood chemistry, blood routine, blood coagulation function and urinalysis indicators 4 days after each injection

SECONDARY OUTCOMES:
Level of S-RBD-specific IgG antibody, titer of neutralizing antibodies, and the number of T cells | from the first vaccination to 12 months after 2 injections
  Evaluate the immunogenicity of ABO1009-DP and ABO-CoV.617.2 against SARS-CoV-2 (original strain, Delta variant and Omicron variant)
Collection of Safety information | through 12 months after 2 injections
  Serious adverse events (SAEs), adverse events of special interest (AESIs) and other medically attended adverse events (MAAEs) through 12 months after 2 injections

CONTACTS AND LOCATIONS:
Overall Officials: Dingfeng Wu, Study Director — Suzhou Abogen Biosciences Co., Ltd.
Locations (2):
- Indonesia (2):
  - Dr. Cipto Mangunkusumo Hospital, Jakarta
  - Persahabatan Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No